CLINICAL TRIAL: NCT06755632
Title: Out-of-hospital Screening of Patients With Significant Hepatic Fibrosis or Cirrhosis and Viral Hepatitis B and C
Brief Title: Screening of Patients With Hepatic Fibrosis or Cirrhosis B and C
Acronym: DEP-CB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APHP240250
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Liver Pathology
Keywords: Cirrhosis, Liver; Hepatic Cirrhosis; Liver Fibrosis; Fibrosis
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Intervention Model Description: screening for liver fibrosis using Fibroscan mini® and will propose rapid diagnostic orientation tests (TROD) for HCV and HBV viral infection, by a traveling physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients of a municipal health center who visit the municipal health center on a given day. (Experimental)
  Interventions: Diagnostic Test: TROD (rapid diagnostic orientation test) and FibroScan®

INTERVENTIONS:
Diagnostic Test: TROD (rapid diagnostic orientation test) and FibroScan® — Fast-track appointment at the hepatology consultation at Avicenne Hospital (Bobigny) or the hepatology consultation at Jean Verdier Hospital (Bondy) for any patient :
  * with Fibroscan® ≥ 9.6 KPa or
  * positive hepatitis C serology or
  * HBsAg positive

SUMMARY:
Regardless of its etiology (chronic hepatitis B or C, alcohol consumption, metabolic steatohepatitis, hemochromatosis, autoimmune liver disease), cirrhosis is a real public health issue. Cirrhosis is a chronic disease and can get complicated by liver cancer, digestive hemorrhage, or liver failure, which are responsible for morbidity and mortality.

In France, cirrhosis prevalence is estimated at 700,000 patients and induce 16,000 deaths per year (10,000 liver cancer and 6,000 liver decompensation). In Ile-de-France area, cirrhosis prevalence is estimated at 130,000 cases, a lot of them are in Seine Saint Denis department due to precariousness.

Hepatitis C virus can now be cured and hepatitis B treatment can suspend hepatitis B replication. All these treatments reduce liver complications but even after virological cure, cirrhosis requires dedicated long term management as well as alcoholic liver disease and metabolic steatohepatitis at cirrhosis stage.

Periodic screening for complications and specific measures were defined by french HAS in 2007 (medication intake, dietary management and specific vaccinations), especially the performance of a semi-annual liver ultrasound for hepatocellular carcinoma (HCC) screening.

Then, it seems essential to screen for patients with viral hepatitis and extensive fibrosis or cirrhosis in our department to achieve active and individualized management of this chronic liver disease, to reduce long term morbidity and mortality.

The main aim of the study is to evaluate the prevalence of advanced liver fibrosis and viral infections B and C in the general population of Seine Saint Denis, using a dual screening method of TROD (rapid diagnostic orientation test) and FibroScan®, combined with a care pathway

DETAILED DESCRIPTION:
Targeted population

The targeted population will be users of one municipal health center visiting the municipal health center on a given day We will propose a screening for liver fibrosis using Fibroscan mini® and will propose rapid diagnostic orientation tests (TROD) for HCV and HBV viral infection, by a traveling physician Expérimental scheme

Proposal by the caregiver to each patient at the center :

* Fibroscan®
* TROD VHC / VHB IF Fibroscan ≥ 9.6 KPa or positive HCV TROD or HBsAg positive THEN Suggested appointment Avicenne hospital hepatology consultation or Jean Verdier hepatology consultation

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Collection of signed consent
* Patients affiliated to a Social Security System

Exclusion Criteria:

* Pregnancy or breastfeeding
* Subjects under AME
* Persons under court protection
* Guardianship or curatorship,
* Safeguard of justice
* Persons under psychiatric care without their consent
* Persons admitted to a health or social institution for purposes other than research,
* Patients of full age under legal protection (guardianship or curatorship)
* Persons unable to express their consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of significant hepatic fibrosis in the general population of Seine Saint Denis | One year of inclusion period

SECONDARY OUTCOMES:
Chronic hepatitis B prevalence | One year of inclusion period
Chronic hepatitis C prevalence | One year of inclusion period
Proportion of eligible patients for management of viral hepatitis B and C | One year of inclusion period
  Proportion of eligible patients for management of viral hepatitis B and C
Prevalence of other causes of chronic liver disease (alcohol and NASH) | One year of inclusion period
Proportion of patients managed in hepatology department after screening for significant fibrosis | One year of inclusion period

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Avicenne Hospital, Bobigny
  - Hepatology department -Hospital Avicenne, Bobigny

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marshall AD, Micallef M, Erratt A, Telenta J, Treloar C, Everingham H, Jones SC, Bath N, How-Chow D, Byrne J, Harvey P, Dunlop A, Jauncey M, Read P, Collie T, Dore GJ, Grebely J. Liver disease knowledge and acceptability of non-invasive liver fibrosis assessment among people who inject drugs in the drug and alcohol setting: The LiveRLife Study. Int J Drug Policy. 2015 Oct;26(10):984-91. doi: 10.1016/j.drugpo.2015.07.002. Epub 2015 Jul 16. PMID 26256938
- [Background] Matthews K, MacGilchrist A, Coulter-Smith M, Jones J, Cetnarskyj R. A nurse-led FibroScan(R) outreach clinic encourages socially deprived heavy drinkers to engage with liver services. J Clin Nurs. 2019 Feb;28(3-4):650-662. doi: 10.1111/jocn.14660. Epub 2018 Sep 24. PMID 30182502
- [Background] Chevaliez S, Pawlotsky JM. New virological tools for screening, diagnosis and monitoring of hepatitis B and C in resource-limited settings. J Hepatol. 2018 Oct;69(4):916-926. doi: 10.1016/j.jhep.2018.05.017. Epub 2018 May 23. PMID 29800630
- [Background] Debette-Gratien M, Francois S, Chevalier C, Alain S, Carrier P, Rigaud C, Abraham B, Burgevin AL, Courat L, Debenes B, Koffi J, Caux-Nussbaum E, Zattoni-Leroy J, Feuillet-Sow G, Dumont Q, Nubukpo P, Loustaud-Ratti V. Towards hepatitis C elimination in France: Scanvir, an effective model to test and treat drug users on dedicated days. J Viral Hepat. 2023 Apr;30(4):355-361. doi: 10.1111/jvh.13798. Epub 2023 Jan 11. PMID 36597183
- [Background] Ganne-Carrie N, Layese R, Bourcier V, Cagnot C, Marcellin P, Guyader D, Pol S, Larrey D, de Ledinghen V, Ouzan D, Zoulim F, Roulot D, Tran A, Bronowicki JP, Zarski JP, Riachi G, Cales P, Peron JM, Alric L, Bourliere M, Mathurin P, Blanc JF, Abergel A, Serfaty L, Mallat A, Grange JD, Attali P, Bacq Y, Wartelle C, Dao T, Benhamou Y, Pilette C, Silvain C, Christidis C, Capron D, Bernard-Chabert B, Zucman D, Di Martino V, Trinchet JC, Nahon P, Roudot-Thoraval F; ANRS CO12 CirVir Study Group. Nomogram for individualized prediction of hepatocellular carcinoma occurrence in hepatitis C virus cirrhosis (ANRS CO12 CirVir). Hepatology. 2016 Oct;64(4):1136-47. doi: 10.1002/hep.28702. Epub 2016 Aug 4. PMID 27348075
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines on non-invasive tests for evaluation of liver disease severity and prognosis - 2021 update. J Hepatol. 2021 Sep;75(3):659-689. doi: 10.1016/j.jhep.2021.05.025. Epub 2021 Jun 21. PMID 34166721